CLINICAL TRIAL: NCT07119164
Title: The Effect of Laughter Yoga Applied to Parents of Mentally Disabled Children on Stress Level, Burnout and Parental Self-Efficacy
Brief Title: Laughter Yoga's Impact on Parental Stress, Burnout, and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Pamukkale University scientific research project department (Unknown)
Responsible Party: Principal Investigator, Burcu Bakırlıoğlu, Research Assistant (PhD Candidate), Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBE-BB-02
Record Dates: First submitted 2025-07-21; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Laughter Yoga; Intellectual Disability; Parents; Burnout; Self Efficacy; Stress
Keywords: Laughter Yoga; Intellectual Disability; Self Efficacy; Parents; Burnout; Stress
MeSH Terms: conditions — Intellectual Disability; Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: The study includes one intervention group and one control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Laughter yoga intervention group (Experimental): A total of 32 mothers who met the inclusion criteria comprised the intervention group and received a total of eight laughter yoga sessions. The laughter yoga intervention was delivered by a researcher certified as a laughter yoga instructor. The intervention protocol was developed within a structured program framework, with each session conducted according to standardized and pre-established guidelines. The laughter yoga sessions encompassed clapping and warm-up exercises, diaphragmatic breathing techniques, incorporation of elements fostering childlike joy and playfulness, as well as guided laughter exercises.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): Thirty-two mothers who met the inclusion criteria constituted the control group. No intervention was administered to the control group. Since the laughter yoga sessions were conducted in a closed environment, the risk of transmission through sound and visual contact was prevented.

INTERVENTIONS:
Other: Laughter yoga — Laughter yoga is a mind-body practice that combines unconditional laughter with yogic breathing techniques (known as pranayama). Developed by Dr. Madan Kataria in 1995, the practice is based on the principle that voluntary laughter can provide similar physiological and psychological benefits as spontaneous laughter. It is typically conducted in group sessions involving eye contact, playful behavior, and laughter exercises, which aim to reduce stress, enhance mood, and promote overall well-being.
  Arms: "Laughter yoga intervention group

SUMMARY:
The present study aims to investigate the effects of laughter yoga on stress levels, burnout, and parental self-efficacy among parents of children with intellectual disabilities.

The specific hypotheses of the study are as follows:

Hypothesis 1: The mean salivary cortisol levels of the intervention group will be significantly lower than those of the control group.

Hypothesis 2: The perceived stress levels of the intervention group will be significantly lower than those of the control group.

Hypothesis 3: The parental self-efficacy levels of the intervention group will be significantly higher than those of the control group.

Hypothesis 4: The burnout levels of the intervention group will be significantly lower than those of the control group.

To assess the effectiveness of the laughter yoga intervention, participants in the intervention group will be compared to a control group of parents who also have children with intellectual disabilities but will not receive any form of intervention. The intervention will consist of a total of eight laughter yoga sessions, conducted twice a week over a four-week period.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children enrolled in the school where the study was conducted
* Parents of children diagnosed with moderate to severe intellectual disability
* Parents who are at least literate
* Parents who can speak and understand Turkish
* Parents with no prior experience in laughter yoga

Exclusion Criteria:

* Parents who have undergone abdominal surgery in the past three months, or those with uncontrolled hypertension, glaucoma, hernia, or epilepsy
* Parents diagnosed with endocrine disorders such as Cushing's or Addison's disease
* Parents on continuous medication (e.g., glucocorticoids, antidepressants, insulin, or oral antidiabetics)
* Pregnant parents
* Parents with hearing, vision, speech, or intellectual disabilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
self-efficacy | 4 weeks
  The scale uses a 7-point Likert-type rating system and consists of 17 items. The total score ranges from a minimum of 17 to a maximum of 119. Higher scores indicate higher levels of self-efficacy. The Cronbach's Alpha internal consistency coefficient of the scale was found to be 0.95.
  When examining the findings related to the reliability and validity of the scale, it was found-contrary to the original version-that the scale has a unidimensional structure. It has been determined to be a valid and reliable tool for assessing the parental self-efficacy levels of mothers and fathers of children with moderate to severe intellectual disabilities in Turkey.
burnout | 4 weeks
  The items are rated on a 4-point scale based on how frequently participants experience the emotions described in the items, ranging from 0 ("never") to 4 ("every day"). The scale consists of two subdimensions: Emotional Exhaustion and Personal Accomplishment.
  The Emotional Exhaustion subscale includes 13 items and has a reliability coefficient of 0.80. Higher average scores on this subscale indicate greater levels of burnout. The Personal Accomplishment subscale consists of 8 items, also with a reliability coefficient of 0.80. Unlike the Emotional Exhaustion subscale, lower average scores on the Personal Accomplishment subscale indicate a higher level of experienced burnout.
Perceived stress | 4 weeks
  The internal consistency coefficient of the scale was calculated as 0.84, and the test-retest reliability coefficient was found to be 0.87. The scale consists of 14 items and is rated on a 5-point Likert-type scale. The total score obtained from the sum of the items reflects the respondent's perceived level of stress, with higher scores indicating a higher level of perceived stress.
stress | 4 weeks
  Stress levels were assessed by analyzing salivary cortisol concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Üniversitesi, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No